CLINICAL TRIAL: NCT02240836
Title: Energy Balance and Breast Cancer Aspects-II Study
Brief Title: Energy Balance and Breast Cancer Aspects-II
Acronym: EBBA-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Inger Thune, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014/945-1
Record Dates: First submitted 2014-09-05; First posted 2014-09-16 (Estimated); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: DCIS Grade 3; Stage I Breast Cancer; Stage II Breast Cancer; LCIS, Lobular Carcinoma in Situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention. Exercise (Experimental): The intervention starts 3-4 weeks after surgical treatment. The exercise program is performed in parallel with standard breast cancer treatment, and take place in supervised exercise groups by experienced physiotherapists. The duration of the intervention exercise program is 12 months, and the participants will attend the exercise groups for training 60 minutes twice a week. Additionally, they will exercise at home for at least 120 minutes a week, aiming to perform a total of 240 minutes of exercise per week
  Interventions: Other: Intervention. Exercise
- Control group (No Intervention): Control group, standard treatment regimen

INTERVENTIONS:
Other: Intervention. Exercise — Physical activity. Attendance in exercise groups 60 min. twice a week and exercise at home 120 min per week. Intervention for 12 months.
  Other Names: Physical activity
  Arms: Intervention. Exercise

SUMMARY:
The purpose of this study, the EBBA-II trial, is to determine whether a 12 month exercise program comprised of strength and endurance training among newly diagnosed breast cancer patients undergoing adjuvant therapy, will influence cardiopulmonary function. Secondary aims are to determine whether the 12 month exercise program will influence factors associated with metabolic profile, tumor growth, disease-free survival, overall mortality and breast cancer specific mortality. Furthermore, the effect on QoL parameters, and dietary factors will be assessed and evaluated.

DETAILED DESCRIPTION:
The EBBA (Energy Balance and Breast cancer Aspects)-II study is a randomized clinical 12 month physical activity intervention trial, including female breast cancer patients diagnosed with histologically verified invasive cancer stage I-II or carcinoma in situ (DCIS/LCIS) grade 3.

* Participants are randomized to either control or intervention group 10 days +/- 2 days after surgery. The intervention start 3 weeks after surgery and continue throughout adjuvant treatments given (chemotherapy, radiation, endocrine therapy etc). The intervention group receive a detailed training program based on their own ventilatory maximal oxygen consumption (VO2max) at baseline. They meet for supervised training sessions in groups for 60 minutes x 2/ week during 12 months. In addition, they are informed to exercise at home for at least of total 120 minutes weekly aiming to perform a total of 240 minutes exercise, weekly. The patients in the control group receive standard of care without any restrictions regarding exercise.
* All participants will undergo a series of measurements before surgery, after surgery, 6 months and after the 12 months exercise intervention trial. Clinical measurements will include anthropometric measurements, fasting blood, fecal and urine samples and cardiopulmonary exercise test (CPET). Complete questionnaires (food diary (PFD)/food frequency questionnaires (FFQ), quality of life (QoL)).
* All participants will come to clinical examination and fasting blood sampling after 2, 3, 5 and 10 years follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Newly diagnosed DCIS grade 3 or invasive breast cancer stage I, II, histologically verified.
* All ethnic groups, but participants have to speak and write the Norwegian language.
* Ability to join and maintain an intervention for 12 months

Exclusion Criteria:

* Verified heart disease
* Dysregulated diabetes mellitus or thyroid disorders
* Muscular and skeletal or other disorders excluding regular physical activity performance
* Body Mass Index >40 kg/m2
* Previous surgical treatment for obesity
* Travel distance >1.5 hour from home to study site

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
VO2max | Baseline,12 months
  Change in VO2max from baseline to 12 months

SECONDARY OUTCOMES:
BMI | Baseline,12 months
  Change in BMI from baseline to 12 months
Systolic blood pressure | Baseline,12 months
  Change in systolic blood pressure from baseline to 12 months
Diastolic blood pressure | Baseline,12 months
  Change in diastolic blood pressure from baseline to 12 months
Total cholesterol | Baseline,12 months
  Change in total cholesterol from baseline to 12 months
LDL cholesterol | Baseline,12 months
  Change in LDL cholesterol from baseline to 12 months
HDL cholesterol | Baseline,12 months
  Change in HDL cholesterol from baseline to 12 months
Total cholesterol/HDL cholesterol | Baseline,12 months
  Change in total cholesterol/HDL cholesterol from baseline to 12 months
HbA1c | Baseline,12 months
  Change in concentrations of HbA1c from baseline to 12 months
Insulin | Baseline,12 months
  Change in concentrations of blood insulin levels (µIU/mL) from baseline to 12 months
Triglycerides | Baseline,12 months
  Change in concentrations of triglycerides from baseline to 12 months
C-reactive Protein (CRP) | Baseline,12 months
  Change in concentrations of CRP (mg/L) from baseline to 12 months
Heart rate | Baseline,12 months
  Change in heart rate from baseline to 12 months
Total fat | Baseline,12 months
  Change in total fat from baseline to 12 months
Truncated fat | Baseline,12 months
  Change in truncated fat from baseline to 12 months
Waist circumference | Baseline,12 months
  Change in waist circumference from baseline to 12 months
Energy from food diary | Baseline,12 months
  Change in energy from food diary from baseline to 12 months
Metabolic syndrome | 12 months
  Dichotomous outcome (yes/no)

OTHER OUTCOMES:
Respiratory Quotient (RQ) | 12 months
  Ratio between the amount of CO2 produced in metabolism and O2 used
Lactate | 12 months
  Blood lactate from fingertip one minute after test
HRmax | 12 months
  Maximal heart rate
BORGmax | 12 months
  Subjective measure of exhaustion
Disease-free survival | Baseline, 1 year, 2 years, 5 years, 10 years
  Time from baseline to the date of cancer symptoms or death
Overall mortality | Baseline, 1 year, 2 years, 5 years, 10 years
  Time from baseline until the date of death, regardless of the cause of death
Breast cancer-specific mortality | Baseline, 1 year, 2 years, 5 years, 10 years
  Time from baseline until the date of breast cancer-specific death
Other exploratory | 12 months
  Forced expiratory volume in 1 second (FEV1), peak expiratory flow (PEF), diffusing capacity of the lung for carbon monoxide (DLco)
  Inflammatory markers, prothrombotic markers, urinary markers, adipokines
  Levels of sex steroid hormones
  Growth factors (Insulin-like growth factor [IGF], insulin, insulin-like growth factor binding protein [IGFBP])
  Microenvironment of the breast, tumor infiltrating lymphocytes (TILS), Crown like structures (CLS)
  Microbiota
  Quality of life and dietary factors

CONTACTS AND LOCATIONS:
Overall Officials: Inger Thune, MD. PhD, Principal Investigator — The Department of Oncology, Ullevål, Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - St. Olavs Hospital, Trondheim

REFERENCES:
- [Background] Thune I, Njolstad I, Lochen ML, Forde OH. Physical activity improves the metabolic risk profiles in men and women: the Tromso Study. Arch Intern Med. 1998 Aug 10-24;158(15):1633-40. doi: 10.1001/archinte.158.15.1633. PMID 9701097
- [Background] Irwin ML, Yasui Y, Ulrich CM, Bowen D, Rudolph RE, Schwartz RS, Yukawa M, Aiello E, Potter JD, McTiernan A. Effect of exercise on total and intra-abdominal body fat in postmenopausal women: a randomized controlled trial. JAMA. 2003 Jan 15;289(3):323-30. doi: 10.1001/jama.289.3.323. PMID 12525233
- [Background] Furberg AS, Veierod MB, Wilsgaard T, Bernstein L, Thune I. Serum high-density lipoprotein cholesterol, metabolic profile, and breast cancer risk. J Natl Cancer Inst. 2004 Aug 4;96(15):1152-60. doi: 10.1093/jnci/djh216. PMID 15292387
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; American Heart Association; National Heart, Lung, and Blood Institute. Definition of metabolic syndrome: Report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Circulation. 2004 Jan 27;109(3):433-8. doi: 10.1161/01.CIR.0000111245.75752.C6. No abstract available. PMID 14744958
- [Background] Courneya KS, Segal RJ, McKenzie DC, Dong H, Gelmon K, Friedenreich CM, Yasui Y, Reid RD, Crawford JJ, Mackey JR. Effects of exercise during adjuvant chemotherapy on breast cancer outcomes. Med Sci Sports Exerc. 2014 Sep;46(9):1744-51. doi: 10.1249/MSS.0000000000000297. PMID 24633595
- [Background] Friedenreich CM, Woolcott CG, McTiernan A, Ballard-Barbash R, Brant RF, Stanczyk FZ, Terry T, Boyd NF, Yaffe MJ, Irwin ML, Jones CA, Yasui Y, Campbell KL, McNeely ML, Karvinen KH, Wang Q, Courneya KS. Alberta physical activity and breast cancer prevention trial: sex hormone changes in a year-long exercise intervention among postmenopausal women. J Clin Oncol. 2010 Mar 20;28(9):1458-66. doi: 10.1200/JCO.2009.24.9557. Epub 2010 Feb 16. PMID 20159820
- [Background] Courneya KS, McKenzie DC, Mackey JR, Gelmon K, Friedenreich CM, Yasui Y, Reid RD, Vallerand JR, Adams SC, Proulx C, Dolan LB, Wooding E, Segal RJ. Subgroup effects in a randomised trial of different types and doses of exercise during breast cancer chemotherapy. Br J Cancer. 2014 Oct 28;111(9):1718-25. doi: 10.1038/bjc.2014.466. Epub 2014 Aug 21. PMID 25144625
- [Background] Edvardsen E, Hem E, Anderssen SA. End criteria for reaching maximal oxygen uptake must be strict and adjusted to sex and age: a cross-sectional study. PLoS One. 2014 Jan 14;9(1):e85276. doi: 10.1371/journal.pone.0085276. eCollection 2014. PMID 24454832
- [Background] Peel AB, Thomas SM, Dittus K, Jones LW, Lakoski SG. Cardiorespiratory fitness in breast cancer patients: a call for normative values. J Am Heart Assoc. 2014 Jan 13;3(1):e000432. doi: 10.1161/JAHA.113.000432. PMID 24419734

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT02240836/SAP_000.pdf